CLINICAL TRIAL: NCT05450120
Title: Neuromuscular Electrical Stimulation and Functional Rehabilitation Protocol in Critically Ill Patients With SARS-CoV-2 Variants in ICUs With Limited Resources: A Randomized Clinical Trial
Brief Title: Rehabilitation of Critically Ill Patients With SARS-CoV-2 Variants in ICU With Limited Resources
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Jacqueline R F Vianna, PhD in physical therapy, postdoctoral student Department of Physical Therapy, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07351119.2.0000.5381
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: COVID-19; intensive care unit; early mobilization; rehabilitation; electrical stimulation; muscle weakness
MeSH Terms: conditions — COVID-19; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Rehabilitation (Active Comparator): Functional rehabilitation protocol
  Interventions: Other: Functional Rehabilitation
- NMES + Functional Rehabilitation (Experimental): Functional rehabilitation protocol associated with neuromuscular electrical stimulation
  Interventions: Other: Functional Rehabilitation; Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Functional Rehabilitation — Functional rehabilitation protocol
Other: Neuromuscular Electrical Stimulation — Neuromuscular electrical stimulation protocol
  Arms: NMES + Functional Rehabilitation

SUMMARY:
Acute rehabilitation in critically ill patients can improve post-intensive care unit (post-ICU) physical function. Scientific evidence has considered neuromuscular electrical stimulation (NMES) as a promising approach for the early rehabilitation of patients during and/or after ICU.

Neuromuscular electrostimulation can be an alternative form of muscle exercise that helps to gain strength in critically ill patients with COVID -19, due to the severe weakness that patients experience due to longer MV, analgesia and NMB duration. Thus, the general objective of evaluating the effects of an early rehabilitation protocol on the strength and functionality of patients affected by SARS-CoV-2 variants and specifically compare the effectiveness of NMES associated with the functional rehabilitation protocol(FR). Also, describe demographics, clinical status, ICU therapies, mortality estimates and Hospital outcomes, of every patients admitted in ICU during the observation periods.

DETAILED DESCRIPTION:
Patients in both groups received the functional rehabilitation protocol adapted from the precoce mobilization protocol of Morris et al, 2008. The protocol was defined in 5 stages, with a period between the application of the stages according to the clinical conditions of the patient, in an interval maximum of 24 hours from the beginning of the application of the first stage. The steps included active assisted mobilization exercises, active with Proprioceptive Neuromuscular Facilitation (PNF) method diagonals for upper limbs and bridge exercises, bedside sitting, balance reactions, weight bearing, transfer to an armchair, passive and active orthostatism, static gait and ambulation. The experimental group also received a protocol of neuromuscular electrical stimulation (NMES), applied bilaterally for 30 minutes, using an electrical stimulator with rectangular pulse waves, symmetrical biphasic, applied to the quadriceps femoris and tibialis anterior muscle at the best motor point, activating fast fibers with a pulse time of less than 300 ms and slow pulses with a pulse time of more than 300 ms, with intensity adjusted to obtain visible muscle contraction and/or according to the patient's tolerance.

ELIGIBILITY:
Inclusion Criteria:

Subjects admitted in ICU for >72hs, undergoing orotracheal intubation and on mechanical ventilation for >48hs, with a diagnosis of Acute Respiratory Distress Syndrome (ARDS) according to Berlin definition secondary to COVID-19, with shock or organ failure, according to the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (7th Interim Edition) Guideline, and clinical stability:

* mean arterial pressure < 60 mmHg;
* heart rate >60 and <120 beats/minute;
* respiratory rate <30 breaths/minute;
* oxygen saturation ≥ 92%;
* fraction of inspired oxygen (FiO2) ≤0.6;
* absence of vasopressor dose increase
* absence of dysrhythmia (except for chronic atrial fibrillation);
* controlled sepsis;
* hemoglobin (Hb) > 8g m/d, plaquettes >20.000, Glucemia >70 e <180;
* without NMBs

Exclusion Criteria:

* Patients with movement resistance
* Walking without assistance before the ICU (except using a cane)
* Cognitive impairment before acute illness
* Signs of intracranial hypertension, neuromuscular disease (myasthenia gravis, amyotrophic lateral sclerosis, Guillain-Barré) and stroke; hip fracture, unstable cervical spine, or pathological fracture
* Prior hospitalization (30 days before ICU)
* Readmission to the ICU, within the current hospitalization
* Presence of an implanted cardiac pacemaker or defibrillator, pregnancy, acute myocardial infarction and, for the experimental group (EG), against indications for NMES (deep vein thrombosis, skin lesions, rhabdomyolysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle strength | 5 months
  Improved skeletal muscle strength by modified Medical Research Council (mMRC)
Functional independence | 5 months
  Improved level of functional independence by ICU Mobility Scale (IMS) and Functional Status Score for the ICU (FSS-ICU)

SECONDARY OUTCOMES:
Mechanical ventilation and hospitalization | 5 months
  Mechanical ventilation time, ICU and hospital stay.
Survived and discharged | 5 months
  Proportion of patients who survived and were discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Vianna, Phd, Principal Investigator — UFSCAR; Jamami, Phd, Study Director — UFSCAR
Locations (1):
- Santa Casa de Batatais, Batatais, São Paulo, Brazil

REFERENCES:
- [Background] Dhand UK. Clinical approach to the weak patient in the intensive care unit. Respir Care. 2006 Sep;51(9):1024-40; discussion 1040-1. PMID 16934166
- [Background] Latronico N, Peli E, Botteri M. Critical illness myopathy and neuropathy. Curr Opin Crit Care. 2005 Apr;11(2):126-32. doi: 10.1097/01.ccx.0000155357.24360.89. PMID 15758592
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Herridge MS. Legacy of intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37(10 Suppl):S457-61. doi: 10.1097/CCM.0b013e3181b6f35c. PMID 20046135
- [Background] De Jonghe B, Sharshar T, Hopkinson N, Outin H. Paresis following mechanical ventilation. Curr Opin Crit Care. 2004 Feb;10(1):47-52. doi: 10.1097/00075198-200402000-00008. PMID 15166849
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Latronico N, Bolton CF. Critical illness polyneuropathy and myopathy: a major cause of muscle weakness and paralysis. Lancet Neurol. 2011 Oct;10(10):931-41. doi: 10.1016/S1474-4422(11)70178-8. PMID 21939902
- [Background] Latronico N. Critical illness polyneuropathy and myopathy 20 years later. No man's land? No, it is our land! Intensive Care Med. 2016 Nov;42(11):1790-1793. doi: 10.1007/s00134-016-4475-4. Epub 2016 Aug 8. No abstract available. PMID 27502507
- [Background] Bolton CF, Gilbert JJ, Hahn AF, Sibbald WJ. Polyneuropathy in critically ill patients. J Neurol Neurosurg Psychiatry. 1984 Nov;47(11):1223-31. doi: 10.1136/jnnp.47.11.1223. PMID 6094735
- [Background] Bonorino KC, Cani KC. Early mobilization in the time of COVID-19. Rev Bras Ter Intensiva. 2020 Oct-Dec;32(4):484-486. doi: 10.5935/0103-507X.20200086. No abstract available. PMID 33470350
- [Background] Hodgson C, Needham D, Haines K, Bailey M, Ward A, Harrold M, Young P, Zanni J, Buhr H, Higgins A, Presneill J, Berney S. Feasibility and inter-rater reliability of the ICU Mobility Scale. Heart Lung. 2014 Jan-Feb;43(1):19-24. doi: 10.1016/j.hrtlng.2013.11.003. Epub 2013 Nov 19. PMID 24373338
- [Background] Zanni JM, Korupolu R, Fan E, Pradhan P, Janjua K, Palmer JB, Brower RG, Needham DM. Rehabilitation therapy and outcomes in acute respiratory failure: an observational pilot project. J Crit Care. 2010 Jun;25(2):254-62. doi: 10.1016/j.jcrc.2009.10.010. Epub 2009 Nov 26. PMID 19942399
- [Background] Bailey PP, Miller RR 3rd, Clemmer TP. Culture of early mobility in mechanically ventilated patients. Crit Care Med. 2009 Oct;37(10 Suppl):S429-35. doi: 10.1097/CCM.0b013e3181b6e227. PMID 20046131
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] Stiller K. Physiotherapy in intensive care: towards an evidence-based practice. Chest. 2000 Dec;118(6):1801-13. doi: 10.1378/chest.118.6.1801. No abstract available. PMID 11115476
- [Background] Maffiuletti NA, Gondin J, Place N, Stevens-Lapsley J, Vivodtzev I, Minetto MA. Clinical Use of Neuromuscular Electrical Stimulation for Neuromuscular Rehabilitation: What Are We Overlooking? Arch Phys Med Rehabil. 2018 Apr;99(4):806-812. doi: 10.1016/j.apmr.2017.10.028. Epub 2017 Dec 9. PMID 29233625
- [Background] De Jonghe, B., Sharshar, T., Lefaucheur, J.-P., & Outin, H. Critical Illness Neuromyopathy. Clinical Pulmonary Medicine. 2005; 12(2): 90-96.
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Result] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Result] Needham DM. Mobilizing patients in the intensive care unit: improving neuromuscular weakness and physical function. JAMA. 2008 Oct 8;300(14):1685-90. doi: 10.1001/jama.300.14.1685. PMID 18840842
- [Result] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Result] Bourdin G, Barbier J, Burle JF, Durante G, Passant S, Vincent B, Badet M, Bayle F, Richard JC, Guerin C. The feasibility of early physical activity in intensive care unit patients: a prospective observational one-center study. Respir Care. 2010 Apr;55(4):400-7. PMID 20406506
- [Result] Maffiuletti NA, Roig M, Karatzanos E, Nanas S. Neuromuscular electrical stimulation for preventing skeletal-muscle weakness and wasting in critically ill patients: a systematic review. BMC Med. 2013 May 23;11:137. doi: 10.1186/1741-7015-11-137. PMID 23701811